CLINICAL TRIAL: NCT03845777
Title: Effects of Iodine-containing Antiseptics on Urine Iodine Levels of Surgical Staff
Brief Title: Urine Iodine Levels of Surgical Staff
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, Assoc. Prof., Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: Capa Iyot
Record Dates: First submitted 2019-02-16; First posted 2019-02-19 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Urine Iodine
Keywords: Iodine; Surgical; Staff; Antiseptic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical Staff: The surgical staff group is the only group of the study. Blood samples of the surgical staff before and after the using antiseptics solution that include iodine were analyzed.
  Interventions: Diagnostic Test: Using Antiseptic solution

INTERVENTIONS:
Diagnostic Test: Using Antiseptic solution — Using of iodine including antiseptic solutions. The investigators investigate the urine iodine status of staff before and after the using of antiseptic solution

SUMMARY:
Objective: The routine use of topical iodinated antiseptic could be a possible cause of iodine contamination. The aim of this study is to evaluate iodine concentrations in operation-room staff who routinely use iodine-containing antiseptics for cleansing of the hands after salt iodization.

Methods: The study included 40 surgeons and surgical nurses who use surgical hand-scrub solutions. Participants applied an iodized brush for a minimum of three times a day on weekdays and were iodine-free on the weekends. Morning spot urine specimens were collected from all participants to analyze the urinary iodine concentration (UIC) twice a week.

DETAILED DESCRIPTION:
Iodine is a major component of thyroid hormones. The recommended dietary allowance for adults is 150 µg per day. Measurement of the urinary iodine concentration (UIC) has been recommended to evaluate the daily nutritional intake of iodine.

According to the 2007 guidelines of the World Health Organization (WHO), the median UIC should be in the range of 100-199 µg/L for adequate daily iodine intake. Before iodization, the use of iodinated antiseptics by operating room staff provided only adequate iodine levels (125 μg/L) and did not lead to toxic doses. When iodization of table salt became mandatory in Turkey in 1998, the median UIC increased to 87 μg/L in 2001, 117 μg/L in 2004, and 130 μg/L in 2007, suggesting sufficient median iodine intake in the general population of Turkey.

In a previous study, the median UIC reached 167 μg/L at least 13 years after iodization, which suggested that iodine prophylaxis is sufficient in Istanbul. However, as a result of the widespread use of amiodarone and iodinated radiological contrast agents in clinical practice, humans are exposed to high doses of exogenous iodine. Furthermore, most surgical hand-scrub solutions contain large amounts of iodine, and transcutaneous and mucosal absorption of iodine from these solutions has been demonstrated. Therefore, the routine use of topical iodinated antiseptic could be a possible cause of iodine contamination after iodization. However, the results of iodine absorption from topical iodine-containing antiseptics are contradictory in several studies. The aim of this study is to reevaluate iodine concentrations in operation-room staff who routinely used iodine-containing antiseptics for cleansing of the hands after a long period of iodization.

MATERIALS AND METHODS This study was carried out between November 2017 and February 2018 with the operating-room staff of Istanbul University Faculty of Medicine. The study included 40 surgeons and surgical nurses who routinely use iodine-containing surgical hand brushes (Surgical Hand Brush Impregnated with 7.5% povidone-iodine). Participants applied the iodized brush for a minimum of three times a day for 3-5 minutes. The exclusion criteria were the use of intravenous iodinated contrast, the use of iodized medications, the use of thyroid hormone replacement, and salt restrictions. The study protocol was approved by the University Hospital Ethics Committee for Human Studies (No: 2017/1127). All volunteer participants provided written informed consent. The subjects used iodine-containing hand scrub solutions on weekdays and were iodine-free on the weekends. Early-morning spot urine specimens were collected from all participants to analyze the UIC twice a week: once at the beginning of the working period (the washout period of the antiseptic) and once at the end of the working period (the antiseptic exposure period). Urine samples were collected in deionized test tubes with tight lids and were immediately transported to the laboratory, acidified, and stored at -80 ºC until analysis.

UICs were determined using the Modified Microplate Method for the Determination of Urinary Iodine Concentration recommended by the CDC's Ensuring the Quality of Urinary Iodine Procedures (EQUIP) booklet with minor modifications as described by Tang et al (CDC, 2011), (Tang et al, 2015). Briefly, urine samples were dissolved at room temperature and incubated with ammonium persulfate (0.9 M final concentration) at 95 ºC on a thermal cycler for 30 minutes. After cooling, 50 µl of digested urine samples were pipetted into microplate wells. 100 µl of 0.05 M arsenious acid solution was added to each well and mixed. Finally, 50 µl of 0.019 M ceric ammonium sulfate solution was added to each well. After incubation for 30 minutes at 25 °C, absorbance at 405 nm was recorded. UICs were determined using a standard curve and expressed in μg/l.

For internal quality control analysis, urine pools (high level: 350 μg/l, low level: 80 μg/l) were prepared from patient samples, portioned, and stored at -80°C. Two levels of pooled urine samples were included in each run for quality control. Between-run coefficients of variation (CV%) for urine iodine measurements were 8.65% for the low level and 11.1% for the high level. Values of 50-99 μg/L were defined as mild iodine deficiency, values of 20-49 μg/L were defined as moderate deficiency, and values < 20 μg/L were defined as severe deficiency. Values of 100-199 μg/L were defined as adequate iodine intake, values of 200-299 μg/L were defined as exceeding iodine requirements, and values ≥ 300 μg/L were defined as potentially harmful to healthy thyroid function.

ELIGIBILITY:
Inclusion Criteria:

* Surgical staff

Exclusion Criteria:

* goiter
* hypertension
* thyroidectomy history

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The surgical staff used iodine-containing hand scrub solutions for antisepsis
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Urine Iodine | 1 week
  The subjects used iodine-containing hand scrub solutions on weekdays and were iodine-free on the weekends. Early-morning spot urine specimens were collected from all participants to analyze the UIC twice a week: once at the beginning of the working period (the washout period of the antiseptic) and once at the end of the working period (the antiseptic exposure period).

CONTACTS AND LOCATIONS:
Overall Officials: Sema Yarman, Prof., Study Director — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Erdogan MF, Tatar FA, Unluturk U, Cin N, Uysal AR. The effect of scrubbing hands with iodine-containing solutions on urinary iodine concentrations of the operating room staff. Thyroid. 2013 Mar;23(3):342-5. doi: 10.1089/thy.2012.0325. PMID 23234312
- [Result] Grasso L, Maxia PL, Bartalena L, Murtas ML, Taberlet A, Martino E. Iodine contamination in subjects admitted to a general hospital. J Endocrinol Invest. 1992 Apr;15(4):307-8. doi: 10.1007/BF03348739. PMID 1512422
- [Result] Michalaki M, Pylioti A, Loutas V, Mamali I, Markou KB. Absence of differences in urinary iodine excretion and thyroid function tests in operating room staff members using or not using iodine-containing antiseptic solutions. Thyroid. 2013 Dec;23(12):1659-60. doi: 10.1089/thy.2013.0218. Epub 2013 Aug 1. No abstract available. PMID 23724900